CLINICAL TRIAL: NCT02517190
Title: Effects of Repeated Short-term Microgravity During Parabolic Flight Conditions on Neuro-endocrine, Immune and Metabolic Changes
Acronym: COSI@PFC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 12-024
Record Dates: First submitted 2015-07-23; First posted 2015-08-06 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Healthy
Keywords: volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stress response measurements (Other)
  Interventions: Other: Parabolic flight; Other: neuro-endocrine measurements; Other: immunological measurements; Other: cellular energy metabolism measurements

INTERVENTIONS:
Other: Parabolic flight
Other: neuro-endocrine measurements — psychic stress tests, stress hormones: prolactin, cortisol, endo-cannabinoids
Other: immunological measurements — blood cell counts, B2 integrins, cytokines, C-reactive protein
Other: cellular energy metabolism measurements — purines, lactate

SUMMARY:
From previous parabolic flight campaigns completed by our research group investigators gathered data showing important changes in neuro-endocrine and also immunological changes. This experiment now will complete the data set-up obtained during the MARS500 study on how these respective individuals will re-act to highly physically and emotionally challenging situations during a parabolic flight.

This add-on experiment to MARS500 will enable answering to the following questions i) if the stress response systems - when compared for two conditions but in the same individuals - do react uniformly and ii) if those subjects prone to have adequate stress response pattern will show gradually less immune modulation effects.

The understanding of the complex interactions of stress and immunity under chronic and acute stress conditions might help to enable adequate health and immune monitoring and might as well suggest suitable countermeasures for the prevention of the unwanted immunological effects during long-term confinement and space missions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (men or women)
* Aged from 18 to 65
* Affiliated to a Social Security system and, for non-French resident, holding a European Health Insurance Card (EHIC)
* Who accepted to take part in the study
* Who have given their written stated consent
* Who participated in the MARS500 experiment
* Who has passed a medical examination similar to a standard aviation medical examination for private pilot aptitude. There will be no additional test performed for subject selection.

Exclusion Criteria:

* Person who took part in a previous biomedical research protocol, of which exclusion period is not terminated
* Pregnant women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-05; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
neuro-endocrine measurements composite | baseline
  prolactin, cortisol, endo-cannabinoids
immunological measurements composite | baseline
  blood cell counts, B2 integrins, cytokines, C-reactive protein
cellular energy metabolism measurements composite | baseline
  purines, lactate

CONTACTS AND LOCATIONS:
Locations (1):
- Umr Ucbn/Inserm U1075 Comete, Caen, Basse-Normandie, France